CLINICAL TRIAL: NCT04256447
Title: High Dietary Salt Intake in Pediatric Patients With Type 1 Diabetes Mellitus Not Related to Overweight and Obesity
Brief Title: High Salt Intake Unrelated to Obesity in Diabetes
Acronym: Diasalt
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Angela Zanfardino, Medical Doctor, University of Campania Luigi Vanvitelli
Other Study IDs: Diasalt
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 1; Food Habits
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sixty-eight children and adolescents with type 1 diabetes: Sixty-eight children and adolescents aged between 4 and 18 years with type 1 diabetes. Patients with celiac disease, thyroid disease, other autoimmune diseases, concurrent illness, patients with diabetic nephropathy, other renal disease and in therapy with natriuretic drugs were excluded.
  Interventions: Diagnostic Test: Urinary sodium concentrations

INTERVENTIONS:
Diagnostic Test: Urinary sodium concentrations — The urinary sodium excretion was measured using an immunochemical methodology

SUMMARY:
People around the world are consuming much more sodium than is physiologically necessary. A number of studies suggest that dietary sodium intake is related to weight gain. The aim of our study was to evaluate in a population of children and adolescents with type 1 diabetes mellitus, possible correlations between the urinary sodium excretion (UNa24h), indirect marker of sodium intake, and both duration of diabetes and BMI z-score(Body Mass Index). Moreover, we also evaluated the correlation between UNa24h and duration of diabetes according with the presence/absence of overweight/obesity.

DETAILED DESCRIPTION:
Elevated sodium intake has been associated with hypertension, cardiovascular diseases and stroke, and decreasing sodium intake may reduce blood pressure and the risk of cardiovascular diseases (CVDs), leading cause of death in the world.

Recent data on sodium intake show that populations around the world are consuming much more sodium than is physiologically necessary.

Studies in children have reported positive associations between sodium intake and adiposity.

The aim of our study was to evaluate in a population of children and adolescents with type 1 diabetes mellitus, possible correlations between the urinary sodium excretion (UNa24h), indirect marker of sodium intake, and both duration of diabetes and BMI z-score. Moreover we also evaluated the correlation between UNa24h and duration of diabetes according with the presence/absence of overweight/obesity.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus

Exclusion Criteria:

* Patients with celiac disease, thyroid disease, other autoimmune diseases, concurrent illness, patients with diabetic nephropathy, other renal disease and in therapy with natriuretic drugs

Ages: 4 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and adolescents affected by type 1 diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Urinary sodium concentrations | three days
  Tested in three 24 h urine samples (immunochemical methodology )

CONTACTS AND LOCATIONS:
Overall Officials: Angela Zanfardino, MD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Centro di Diabetologia Pediatrica "G.Stoppoloni", Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Campanozzi A, Avallone S, Barbato A, Iacone R, Russo O, De Filippo G, D'Angelo G, Pensabene L, Malamisura B, Cecere G, Micillo M, Francavilla R, Tetro A, Lombardi G, Tonelli L, Castellucci G, Ferraro L, Di Biase R, Lezo A, Salvatore S, Paoletti S, Siani A, Galeone D, Strazzullo P; MINISAL-GIRCSI Program Study Group. High sodium and low potassium intake among Italian children: relationship with age, body mass and blood pressure. PLoS One. 2015 Apr 8;10(4):e0121183. doi: 10.1371/journal.pone.0121183. eCollection 2015. PMID 25853242
- [Result] Lucko AM, Doktorchik C, Woodward M, Cogswell M, Neal B, Rabi D, Anderson C, He FJ, MacGregor GA, L'Abbe M, Arcand J, Whelton PK, McLean R, Campbell NRC; TRUE Consortium. Percentage of ingested sodium excreted in 24-hour urine collections: A systematic review and meta-analysis. J Clin Hypertens (Greenwich). 2018 Sep;20(9):1220-1229. doi: 10.1111/jch.13353. Epub 2018 Aug 12. No abstract available. PMID 30101426
- [Result] Geserick M, Vogel M, Gausche R, Lipek T, Spielau U, Keller E, Pfaffle R, Kiess W, Korner A. Acceleration of BMI in Early Childhood and Risk of Sustained Obesity. N Engl J Med. 2018 Oct 4;379(14):1303-1312. doi: 10.1056/NEJMoa1803527. PMID 30281992